CLINICAL TRIAL: NCT03604874
Title: High Dose Versus Low Dose Oxytocin for Augmentation of Delayed Labour in Obese Women: A Randomized Clinical Trial
Brief Title: High Dose Versus Low Dose Oxytocin for Augmentation of Delayed Labour in Obese Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OBOX
Record Dates: First submitted 2018-07-21; First posted 2018-07-30 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: DELAYED LABOUR
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low dose oxytocin (Active Comparator): patients will receive intravenous infusion of 5 Units of oxytocin/500 mL lactated ringer solution. Starting rate will be 2 mU/min, incrementally increase by 2 mU/min every 30 minutes until achievement of adequate uterine contractions.
  Interventions: Drug: Oxytocin
- high dose oxytocin (Experimental): patients will receive intravenous infusion of 5 Units of oxytocin/500 mL lactated ringer solution. Starting rate will be 4 mU/min, incrementally increase by 4 mU/min every 30 minutes until achievement of adequate uterine contractions
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — intravenous infusion

SUMMARY:
Obesity is one of the biggest public health problems of the 21st century as it increases the risk of many co-morbid medical conditions. Obesity in pregnancy places women at higher risk of obstetrical complications during pregnancy, delivery and puerperium. Obesity is a risk factor for cesarean delivery, failed induction of labor and labor dystocia, and prolonged labor curves especially among women with class III obesity.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous onset of labor.
* Body mass index ≥ 30 kg/m2.
* Gestational age ≥ 37 weeks.
* Singleton pregnancy.
* Cephalic presentation.
* Reassuring fetal heart rate monitoring.
* Inefficient uterine contractions during active labor
* Women who will accept to participate in the study.

Exclusion Criteria:

* Non-reassuring fetal assessment at the time of recruitment.
* Women received cervical ripening agents.
* Any patients contraindicated for vaginal delivery.
* Multiple gestations.
* Malpresentation.
* Previous cesarean delivery.
* Patients with cardiac diseases, pre-eclampsia or any other medical disorders.
* Fetal demise.
* Intrauterine growth restriction.
* Estimated fetal weight ≥ 5000 grams.
* Pre-labor rupture of membranes > 24 hours.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
The mean duration from oxytocin augmentation initiation to delivery | 12 hours
  the calculated time between oxytocin infusion till delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No